CLINICAL TRIAL: NCT07392255
Title: A First in Human Phase 1 / 2 Multi-center Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of CTx001 Administered Via a Single Subretinal Injection in Patients With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: An Optimised GA Interventional Trial (Opti-GAIN) to Test if Treatment With CTx001 is Safe and Works for People With Geographic Atrophy (GA)
Acronym: Opti-GAIN
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Complement Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTx001-01
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Geographic Atrophy Secondary to Age-related Macular Degeneration
MeSH Terms: interventions — exagamglogene autotemcel

STUDY DESIGN:
Intervention Model Description: Part 1 is a multi-center, open-label, dose-escalation study of 3 doses in 3 cohorts (Cohorts 1 to 3).
  Part 2 is a multi-center, open-label, dose-expansion study in 2 cohorts (Cohorts 4 and 5)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Low Dose
  Interventions: Genetic: CTx001
- Cohort 2 (Experimental): Medium Dose
  Interventions: Genetic: CTx001
- Cohort 3 (Experimental): High Dose
  Interventions: Genetic: CTx001
- Cohort 4 (Experimental): Expansion of a dose selected from Cohort 1-3
  Interventions: Genetic: CTx001
- Cohort 5 (Experimental): Expansion of a second dose selected from Cohort 1-3
  Interventions: Genetic: CTx001

INTERVENTIONS:
Genetic: CTx001 — Subretinal administration of CTx001

SUMMARY:
This is a clinical study to evaluate the safety, tolerability and efficacy of CTx001, administered via a single subretinal injection, for GA (secondary to AMD).

Safety and efficacy will be measured at regular intervals for 2 years after which long-term safety will be assessed annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

Meet protocol-defined age eligibility

Have bilateral geographic atrophy secondary to AMD, confirmed by the Reading Center

Meet baseline lesion size requirements, as assessed by fundus autofluorescence imaging

Meet best-corrected visual acuity and low-luminance visual acuity criteria, as measured by ETDRS charts

Meet retinal sensitivity criteria, as measured by microperimetry

Have sufficient fellow-eye visual function to ensure navigational vision

Have adequate historical SD-OCT imaging available for longitudinal assessment

Meet reproductive status and contraception requirements, where applicable

Be able and willing to provide informed consent and comply with study procedures

Exclusion Criteria:

Macular atrophy or retinal disease not attributable to AMD

Evidence of current or prior choroidal neovascularization (wet AMD)

Prior intraocular, macular, or retinal surgery or laser treatment that may confound assessments

Prior AMD-directed or intravitreal therapy in the study eye, except permitted supplements

Prior exposure to complement inhibitor therapies

Ocular conditions, infections, inflammation, or media opacities that interfere with safety or retinal imaging

Uncontrolled glaucoma, diabetic retinopathy, or clinically significant refractive error

Aphakia or compromised posterior capsule, except as permitted by protocol

Systemic medical or psychiatric conditions that may increase risk or limit compliance

Recent participation in another interventional clinical study or exposure to investigational therapies

Any condition that, in the investigator's judgment, poses unacceptable risk or precludes safe participation

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
To monitor the safety and tolerability of a single administration of CTx001 at 3 dose levels | From dosage to Week 52
  Incidence and severity of ocular and non-ocular adverse events (AE)s and serious AEs (SAEs) up to Week 52 (Year 1)

SECONDARY OUTCOMES:
To evaluate the preliminary efficacy of treatment with CTx001 through changes in the structural and functional parameters of geographic atrophy (GA) | From dosage to Year 1
  Change from baseline in the rate of total ellipsoid zone (EZ) attenuation as measured by spectral domain-optical coherence tomography (SD-OCT) at Week 52 (Year 1)
To evaluate the preliminary efficacy of treatment with CTx001 through changes in the structural and functional parameters of geographic atrophy (GA) | From dosage to Year 1
  Rate of change from baseline in sensitivity as measured by microperimetry at Week 52 (Year 1)
To evaluate the preliminary efficacy of treatment with CTx001 through changes in the structural and functional parameters of geographic atrophy (GA) | From dosage to Year 1
  Change from baseline in low luminance visual acuity (LLVA) as measured by Early Treatment Diabetic Retinopathy Study (EDTRS) chart and neutral density filter at Week 52 (Year 1)
To evaluate the preliminary efficacy of treatment with CTx001 through changes in the structural and functional parameters of geographic atrophy (GA) | From dosage to Year 2
  Change from baseline in the rate of enlargement of lesion area of geographic atrophy as measured by Fundus Auto Fluorescence (FAF) at Week 104 (Year 2)
To evaluate the preliminary efficacy of treatment with CTx001 through changes in the structural and functional parameters of geographic atrophy (GA) | From dosage to Year 2
  Change from baseline in best corrected visual acuity (BCVA) as measured by Early Treatment Diabetic Retinopathy Study (EDTRS) chart at Week 104 (Year 2)
To monitor the long-term safety and tolerability of a single administration of CTx001 at 3 dose levels | From dosage up to Week 260 (Year 5)
  * Incidence and severity of ocular and non-ocular AEs and SAEs up to Week 260 (Year 5)
  * Incidence and extent of retinal pigmentary changes up to Week 260 (Year 5)
To assess immunogenicity to adeno-associated virus Serotype 2 (AAV2)-vector and mini-CR1 transgene product | From dosage up to Week 260 (Year 5)
  Measurement of systemic antibody levels to AAV2-vector and mini-CR1 transgene up to Week 260 (Year 5)

CONTACTS AND LOCATIONS:
Locations (1):
- Sierra Eye Associates, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No